CLINICAL TRIAL: NCT00526214
Title: Multi-center, Prospective Randomized, Comparative Open With Blinded Endpoints (PROBE) Trial to Assess the Safety and Effectiveness of Administration of Celecoxib in Patients With Intracerebral Hemorrhage
Brief Title: Administration of Celecoxib for Treatment of Intracerebral Hemorrhage : A Pilot Study
Acronym: ACE-ICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-0704-028-205; 12-2007-0084
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2010-03

CONDITIONS: Intracerebral Hemorrhage
Keywords: Spontaneous intracerebral hemorrhage; Acute Spontaneous, Supratentorial intracerebral hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): In the control group, patients will not take the drug. We do not use placebo drugs.
- 2 (Experimental): In the intervention group, patients will take celecoxib.
  Interventions: Drug: celecoxib medication

INTERVENTIONS:
Drug: celecoxib medication — In the celecoxib group, patients will take celecoxib 400mg twice (per day), orally for 14 days.
  Other Names: celecoxib(celebrex)
  Arms: 2

SUMMARY:
Primary:

Change of volume of perihematomal edema as assessed by brain CT.

Secondary:

The change of ICH volume between the initial and the follow-up CT scans The neurological status at 90 day using E-GOS and mRS. The cumulative incidence of major and minor adverse events that occurred during and after hospitalization until the end of the study

DETAILED DESCRIPTION:
1. INCLUSION/EXCLUSION CRITERIA

   1. Inclusion Criteria

      * Spontaneous intracerebral hemorrhage was documented by CT scanning within 24 hours of the onset of symptoms
      * Supratentorial location of hemorrhage
      * Older than 17 yrs
      * Informed consent before study
   2. Exclusion Criteria

      * Planned surgical evacuation of hematoma within 24hrs
      * Secondary ICH such as trauma or aneurysmal rupture
      * Taking anticoagulation previously
      * Pregnancy,known allergy to celecoxib, severe liver or kidney disease, or poor performance state were excluded
      * Other physical condition, making the patient difficult to participate in this study (decided by the neurologist or the physician).
2. OTHER THERAPY

   -No limitation of other medications except NSAIDs, anticoagulation and antiplatelet agent because of aggravating the symptoms
3. STUDY DESIGN Multicenter, prospective randomized, comparative open with blinded endpoints (PROBE) trial to assess the safety and effectiveness of administration of celecoxib for 14 days in patients with intracerebral hemorrhage

ELIGIBILITY:
Inclusion Criteria:

1. Spontaneous intracerebral hemorrhage was documented by CT scanning within 24 hours of the onset of symptoms
2. Supratentorial location of hemorrhage
3. Older than 17 yrs

Exclusion Criteria:

1. Planned surgical evacuation of hematoma within 24hrs
2. Secondary ICH due to trauma or aneurismal rupture or etc
3. Taking antithrombotics or other NSAIDs previously
4. Pregnancy
5. Other physical condition, making the patient difficult to participate the study (decided by the neurologist or the physician).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change of volume of perihematomal edema as assessed by brain CT | at 1st day of admission and repeated at 7th±1 day
  Brain CT scanning for measurement of volumes of ICH and perihematomal edema was performed at 1st day of admission and repeated at 7th±1 day. Considering some possible errors in measurement of edema volume, at follow-up CT scan, the decrease more than 20% from the initial edema volume was coded as "decreased" edema volume; the increase more than 20% was coded as "increased"; the change between -20% and 20% was coded as "unchanged".

SECONDARY OUTCOMES:
The neurological status at 90 day using E-GOS and mRS | 90 days after onset.
  The secondary endpoints were neurological status at 90 day using E-GOS and mRS. Good outcome was defined as 6 or more in E-GOS score, and 2 or less in mRS score.
Change of ICH volume between the initial and the follow-up CT scans | Day1, Day 7
  Change of ICH volume between the initial and the follow-up CT scans. In this analysis, the 20% criterion was applied as mentioned in the edema analysis
Major and minor adverse events | anytime for 3 months
  the cumulative incidence of major and minor adverse events that occurred during and after hospitalization until the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Kyu Roh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Chu K, Jeong SW, Jung KH, Han SY, Lee ST, Kim M, Roh JK. Celecoxib induces functional recovery after intracerebral hemorrhage with reduction of brain edema and perihematomal cell death. J Cereb Blood Flow Metab. 2004 Aug;24(8):926-33. doi: 10.1097/01.WCB.0000130866.25040.7D. PMID 15362723